CLINICAL TRIAL: NCT05338671
Title: Effect of Post-Operative Anesthetics on Post-Operative Pain in Patients Receiving Endodontic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Avina Paranjpe, Professor: School of Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00013406
Record Dates: First submitted 2021-06-19; First posted 2022-04-21 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Endodontic Disease; Post Operative Pain; Symptomatic Irreversible Pulpitis
Keywords: endodontics; root canal; lidocaine; bupivicaine; ibuprofen; symptomatic irreversible pulpitis; post operative pain; heft parker visual analog scale
MeSH Terms: conditions — Dental Pulp Diseases; Pain, Postoperative | interventions — Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: Two different arms each receiving an inferior alveolar nerve block with two different local anesthetics
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2% Lidocaine 1:100,000 epinephrine (Active Comparator): Participants in this arm will receive an inferior alveolar nerve block with 1 cartridge (1.8 mL) of 2% Lidocaine 1:100,000 epinephrine following endodontic treatment.
  Interventions: Drug: Local anesthetic
- 0.5% bupivicaine 1:200,000 epinephrine (Active Comparator): Participants in this arm will receive an inferior alveolar nerve block with 1 cartridge (1.8 mL) of 0.5% bupivicaine 1:200,000 epinephrine following endodontic treatment.
  Interventions: Drug: Local anesthetic

INTERVENTIONS:
Drug: Local anesthetic — Patients will receive inferior alveolar nerve block injection following endodontic treatment.

SUMMARY:
This study will assess the efficacy of two local anesthetics (2% lidocaine 1:100,000 epinephrine and 0.5% bupivicaine 1:200,000 epinephrine) in reducing post-operative pain in patients receiving endodontic treatment.

DETAILED DESCRIPTION:
The goal of this study is to assess the efficacy of 2% lidocaine 1:100,000 epinephrine and 0.5% bupivicaine 1:200,000 epinephrine in reducing post-operative pain in patients with symptomatic irreversible pulpitis on a mandibular tooth that receive endodontic treatment. Participants of this study will include patients that present to the University of Washington Endodontic clinic and fit the inclusion criteria of being >18 years old, healthy (ASA I or II) and having a diagnosis of symptomatic irreversible pulpitis on a mandibular tooth, that is willing to undergo endodontic treatment in two visits. Upon diagnosis, and informed consent, patients will be asked to participate in this study. If enrolled in the study, participants will receive standard endodontic treatment with temporary placement of Calcium Hydroxide medicament within the canals of the tooth and placement of a temporary filling. They will then be randomized to receive an inferior alveolar nerve block with 1 cartridge (1.8mL) of either 2% lidocaine 1:100,000 epinephrine or 0.5% bupivicaine 1:200,000 epinephrine. Patients will be given a form to track their pain levels for the next 72 hours, that they will return at a follow up visit. This form will use the Heft-Parker visual analog pain scale to track pain levels as well as ask participants to track their use of over the counter analgesics, in particular, Advil/ibuprofen. The pain tracking form will be returned to the clinic and root canal will be completed also at this follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic irreversible pulpitis on mandibular, posterior tooth
* ASA I or II
* >18 years old

Exclusion Criteria:

* Maxillary or mandibular anterior tooth
* Diagnosis of pulp necrosis or reversible pulpitis
* Tooth deemed non-restorable
* <18 years old
* ASA III, IV, or V
* Patients who are contraindicated to take ibuprofen
* Patients with allergies to any medications being assessed in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avina Paranjpe, Principal Investigator — University of Washington
Locations (1):
- University of Washington- School of Dentistry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Kahtani A. Effect of long acting local anesthetic on postoperative pain in teeth with irreversible pulpitis: Randomized clinical trial. Saudi Pharm J. 2014 Jan;22(1):39-42. doi: 10.1016/j.jsps.2013.01.004. Epub 2013 Jan 26. PMID 24493972
- [Background] Dunsky JL, Moore PA. Long-acting local anesthetics: a comparison of bupivacaine and etidocaine in endodontics. J Endod. 1984 Sep;10(9):457-60. doi: 10.1016/S0099-2399(84)80270-8. No abstract available. PMID 6387029
- [Background] Moradi S, Naghavi N. Comparison of bupivacaine and lidocaine use for postoperative pain control in endodontics. Iran Endod J. 2010 Winter;5(1):31-5. Epub 2010 Feb 20. PMID 24778680
- [Background] Parirokh M, Yosefi MH, Nakhaee N, Manochehrifar H, Abbott PV, Reza Forghani F. Effect of bupivacaine on postoperative pain for inferior alveolar nerve block anesthesia after single-visit root canal treatment in teeth with irreversible pulpitis. J Endod. 2012 Aug;38(8):1035-9. doi: 10.1016/j.joen.2012.04.012. Epub 2012 May 30. PMID 22794202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine
Started | 18 | 17
Completed | 15 | 15
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Root canal completed in a single visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.1) | 37.2 (17.2) | 38.2 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Level 6 Hours on a Visual Analog Scale
Description: Participants will be asked to track the amount of pain they have following their endodontic treatment using the Heft-Parker visual analog scale with scores ranging from 0-170 with higher scores signifying more pain.
Time Frame: Patients will be asked to track pain levels at 6 post-operatively on a visual analog scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine
Number analyzed (Participants) | 15 | 15
units on a scale | 64.2 (43.9) | 43.1 (43.1)

2. Primary Outcome: Post-operative Pain Level 12 Hours on a Visual Analog Scale
Description: as for outcome 1
Time Frame: Patients will be asked to track pain level at 12 hours post-operatively on a visual analog scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine
Number analyzed (Participants) | 15 | 15
units on a scale | 67.4 (44.9) | 45.1 (34.5)

3. Primary Outcome: Post-operative Pain Level 24 Hours on a Visual Analog Scale
Description: as for outcome 1
Time Frame: Patients will be asked to track pain level at 24 hours post-operatively on a visual analog scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine
Number analyzed (Participants) | 15 | 15
units on a scale | 48.9 (27.9) | 36.5 (32.5)

4. Primary Outcome: Post-operative Pain Level 48 Hours on a Visual Analog Scale
Description: as for outcome 1
Time Frame: Patients will be asked to track pain level at 48 hours post-operatively on a visual analog scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine
Number analyzed (Participants) | 15 | 15
units on a scale | 45.3 (34.1) | 30.1 (34.2)

5. Primary Outcome: Post-operative Pain Level 72 Hours on a Visual Analog Scale
Description: as for outcome 1
Time Frame: Patients will be asked to track pain level at 72 hours post-operatively on a visual analog scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine
Number analyzed (Participants) | 15 | 15
units on a scale | 35.5 (41.6) | 21.9 (26.7)

ADVERSE EVENTS:
Time Frame: Patients were followed up for 72 hours to check for any adverse reactions
Arm/Group | 2% Lidocaine 1:100,000 Epinephrine | 0.5% Bupivicaine 1:200,000 Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

LIMITATIONS AND CAVEATS:
Limitations/future direction

* Sample size
* Lack of a control group: Inferior alveolar nerve block with saline solution
* Lack of inclusion of other pre-operative pulpal diagnoses: Pulp Necrosis, Previously Initiated Therapy, Previously Treated
* Lack of inclusion of maxillary posterior teeth
* We could have tracked patients for longer periods of time to examine persistent pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT05338671/Prot_SAP_000.pdf